CLINICAL TRIAL: NCT05122715
Title: Demonstration Of A Next Generation PET CT System (OMNI dBGO)
Brief Title: Demonstration Of A Next Generation PET CT System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 215514655
Record Dates: First submitted 2021-11-01; First posted 2021-11-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-02

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OMNI PET/CT scan first (Other)
  Interventions: Device: Additional PET/CT Scan
- DMI PET/CT scan first (Other)
  Interventions: Device: Additional PET/CT Scan

INTERVENTIONS:
Device: Additional PET/CT Scan — The subject will undergo two PET/CT scans, one on the DMI scanner and one on the OMNI scanner.

SUMMARY:
The intent of this evaluation is to obtain user feedback on device performance, user preference, image quality, workflow, and new device features, a necessary part of product development. This study will also help to inform protocol development in reducing both scan time and/or radiologic tracer dose. The goal of this study is to collect a library of image data from the hybrid PET/CT system to be used for evaluation and optimization of the image quality of the system in a clinical setting and as comparison with the standard of care hybrid PET/CT system, Discovery MI 25m (DMI5R).

ELIGIBILITY:
Inclusion Criteria:

1. Adult, who is at least 18 years of age;
2. A clinical indication for PET/CT examination according to current clinical practice standards;
3. Able and willing to provide informed consent for participation in this study

Exclusion Criteria:

1. Diabetic patient with a glucose level ≥ 150 mg/dl at the time of the exam (for FDG) or,
2. Known to be pregnant or breastfeeding (the investigational site will follow their standard practice of verifying for women of childbearing age. No study specific pregnancy test will be performed for this study); or,
3. Previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation- Likert Scale | through study completion, an average of 1 year
  The primary endpoints of this study are completed image evaluation using a 1 point Likert Scale of the OMNI PET/CT system including analysis, reading, and scoring utilizing a Likert Scale, by three (3) qualified Nuclear Medicine physicians.

SECONDARY OUTCOMES:
Data Collection | through study completion, an average of 1 year
  PET/CT Image collection

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Thomsen, Study Director — GE Healthcare
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No